CLINICAL TRIAL: NCT06896149
Title: Association Between Mild Fetal Hydronephrosis (G1-G2), Gestational Diabetes and Spontaneous Resolution in the First Year of Life vs Moderate-severe Fetal Hydronephrosis (G3-G4), Obstructive Causes and Worse Postnatal Outcome
Brief Title: Mild Fetal Hydronephrosis, Gestational Diabetes and Spontaneous Resolution vs Moderate-severe Fetal Hydronephrosis, Obstructive Causes and Worse Postnatal Outcome
Acronym: FHYDO
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7077
Record Dates: First submitted 2025-01-29; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-01

CONDITIONS: Hydronephrosis; Gestational Diabetes
MeSH Terms: conditions — Hydronephrosis; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fetal hydronephrosis (cases): * Single pregnancy in normal progression, in presence of single or bilateral fetal hydronephrosis of any grade of severity from G1 to G4 with a gestational diabetes diagnosis (cases).
  * Single pregnancy in normal progression, in presence of single or bilateral fetal hydronephrosis of any grade of severity from G1 to G4 without a gestational diabetes diagnosis (cases).
  Interventions: Diagnostic Test: Obstetric ultrasound
- No fetal hydronephrosis (controls): * Single physiological pregnancy in normal evolution without finding of fetal hydronephrosis and gestational diabetes.
  * Single pregnancy with a diagnosis of gestational diabetes in the absence of fetal hydronephrosis.
  Interventions: Diagnostic Test: Obstetric ultrasound

INTERVENTIONS:
Diagnostic Test: Obstetric ultrasound — Ultrasound focus on fetal renal pelvis, amniotic fluid assessment, and fetal weight estimation.
  Other Names: Data collection of oral glucose tolerance test, fasting blood glucose, or glycated hemoglobin.; Collection of postnatal kidney and urinary tract ultrasound examination data, performed according to clinical protocols, up to 6 months of postnatal life.

SUMMARY:
Renal pelvis dilatation can be a relatively common finding on obstetric antenatal ultrasounds occurring in 1% to 5% of all pregnancies, with a known predilection for the male sex. Fetal hydronephrosis can be ascribed to structural obstructive conditions or functional origin causes. The latter are characterized by the transience of the clinical picture, which appears milder in degree, onset at later gestational ages, a course of substantial stability and spontaneous regression, sometimes as early as during pregnancy or early postnatal life. Fetal hydronephrosis related to structural obstructive causes, on the other hand, classically presents an earlier onset, a worsening course during pregnancy and often requires postnatal surgical correction. Additional ultrasound findings that contribute to prognosis include those indicative of an associated congenital anomaly of the kidneys and urinary tract (CAKUT). The risk of postnatal pathology in mild prenatal hydronephrosis is reported to be between 11% and 15%. It increases up to 27-45% in fetuses with moderate prenatal hydronephrosis and up to 53- 88% in cases of severe hydronephrosis. In the outpatient clinical practice of prenatal ultrasonography, is hypothesized an association between mild, mono- bilateral fetal hydronephrosis as an isolated ultrasound finding and gestational diabetes. In this population, this study aims to highlight the stability of the sonographic picture, relative improvement with effective glycemic control with diet or medical therapy, and subsequent spontaneous resolution in early postnatal life. A possible causal link between the two conditions could lie in the association of poorly controlled gestational diabetes with fetal hyperglycemia, which would cause increased osmotic diuresis resulting in polyuria and subsequent hydronephrosis. In contrast, is hypothesized an association between earlier-onset moderate-to-severe fetal hydronephrosis, its worsening progression throughout pregnancy and the anatomic abnormalities finding in the fetal urinary tract, in no correlation with maternal gestational diabetes. This condition correlates with increased postnatal complications (e.g., recurrent urinary infections, need for antibiotic prophylaxis, etc.) and a more severe postnatal outcome that may require surgical correction. To date, there is limited scientific literature concerning the functional causes of fetal hydronephrosis, as opposed to obstructive causes, which have been more analyzed and classified. This ambispective observational case-control study aims to evaluate pregnant women accessing the obstetric ultrasound and obstetric day hospital outpatient clinics of the Fondazione Policlinico A. Gemelli- IRCCS with ultrasound finding of mono-bilateral fetal hydronephrosis during the second and third trimester of pregnancy. In this population we will define the fetal hydronephrosis degree, its evolution, the association with maternal metabolic disorders, in order to estimate postnatal morbidity. All prenatal ultrasound images will be interpreted by the same group of specialists. To assess the degree of fetal hydronephrosis, the classification system developed by SFU in 1993 will be used. The latter is the most commonly used among pediatric urologists for grading neonatal and infant pelvic disorders:

* grade 0: no dilatation, calico walls paired with each other
* grade 1 (mild): dilation of the renal pelvis without dilation of the calyces
* grade 2 (mild): dilatation of the renal pelvis (mild) and calyces
* grade 3 (moderate): moderate dilatation of the renal pelvis and calyces; dulling of the fornixes and flattening of the papillae; possible mild cortical thinning
* grade 4 (severe): gross dilatation of renal pelvis and calyces; cortical thinning.

The diagnosis of gestational diabetes will be defined by an altered oral glucose tolerance test (OGTT) result or elevated glycosylated hemoglobin (HBA1c) values. In addition, the presence of a flat OGTT trend suggestive of an insulin resistance condition will also be considered pathological. The OGTT will be performed between weeks 24 and 28 of pregnancy, as per the guidelines. In patients at high risk of developing gestational diabetes, early screening will be performed between sixteen and eighteen weeks of pregnancy. Amniotic fluid will be assessed according to one of the following ultrasound criteria:

* calculation of amniotic fluid index (AFI) by summing the vertical depth of amniotic fluid measured in each quadrant of the uterus
* With the single deepest pocket (SDP). Polydramnios is diagnosed when the amniotic fluid index (AFI) is ≥ 250 mm, the single deepest pocket (SDP) is ≥ 80 mm, or when the examiner subjectively assesses an increase in amniotic fluid. Oligohydramnios is diagnosed when the AFI is ≤ 50 mm or when the SDP is ≤ 20 mm.

ELIGIBILITY:
Inclusion criteria

* Written informed consent.
* Single pregnancy in normal progression, in presence of single or bilateral fetal hydronephrosis of any grade of severity with or without a gestational diabetes diagnosis and without evidence of other ultrasound detectable abnormalities of the fetus affecting other anatomical districts (cases).
* Single physiological pregnancy in normal evolution without finding of fetal hydronephrosis and gestational diabetes (controls).
* Single pregnancy with a diagnosis of gestational diabetes in the absence of fetal hydronephrosis (controls).
* Having performed at least one prenatal ultrasound at the obstetric ultrasound clinics and obstetric DH of the Foundation.
* Have been screened for gestational diabetes.

Exclusion Criteria

* Detection of other major malformations and genetic syndromes in the fetus.
* Twin pregnancies.
* Maternal conditions such as diabetes insipidus, type I and type II diabetes mellitus.

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant women accessing the Obstetric ultrasound clinics and the obstetrics DH of Fondazione Policlinico A. Gemelli- IRCCS with or without a diagnosis of gestational diabetes, with ultrasound finding of fetal hydronephrosis of different grades and assessment of the evolution of hydronephrosis in the newborn in the first six months of postnatal life.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Mild fetal Hydronephrosis in patients with gestational diabetes | 1 year
  This study aims to evaluate if gestational diabetes can be associated with mild grade (G1-G2) fetal hydronephrosis based on all clinical data present at the time of admission and obstetric ultrasound data.

SECONDARY OUTCOMES:
Fetal hydronephrosis grade in women with and without gestational diabetes | 3 years
  to compare fetal hydronephrosis in pregnant women with and without gestational diabetes
Moderate to severe fetal hydronephrosis and gestational diabetes | 3 years
  To demonstrate the absence of association between moderate-to-severe fetal hydronephrosis (G3-G4) and gestational diabetes, collecting all clinical data present at the time of admission and obstetric ultrasound data.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Romiti, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, UOC Ostetricia e patologia ostetrica, Roma, Italia, Italy